CLINICAL TRIAL: NCT04248868
Title: Recombinant tPA by Endovascular Administration for the Treatment of Submassive Pulmonary Embolism Using Pharmaco-mechanical Catheter Directed Thrombolysis for the redUction of Thrombus burdEn
Brief Title: tPA by Endovascular Administration for the Treatment of Submassive PE Using CDT for the Reduction of Thrombus Burden
Acronym: RESCUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thrombolex, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THRO-CLIN-2019-01
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Catheter Directed Therapy
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Pulse Spray and Infusion of r-tPA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- BEC Treatment (Experimental): The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery.
  Interventions: Device: The Bashir™ Endovascular Catheter; Drug: r-tPA

INTERVENTIONS:
Device: The Bashir™ Endovascular Catheter — The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature.
Drug: r-tPA — Pulse spray and infusion

SUMMARY:
To demonstrate the efficacy and safety of the Bashir™ Endovascular Catheter for the administration of pharmaco-mechanical catheter directed therapy using low dose r-tPA for the treatment of acute submassive pulmonary embolism.

DETAILED DESCRIPTION:
The Bashir™ Endovascular Catheter has been designed to administer therapeutic agents in the peripheral vasculature. Because of the unique design of the catheter, with its six expandable infusion limbs, the Bashir™ Endovascular Catheter has the ability to: 1. Create a much larger central channel for blood flow, thereby utilizing the body's own endogenous fibrinolytic agents to lyse the clot, and 2. Greatly enhance the radial dispersion of a catheter-administered thrombolytic agent throughout the thrombus. Expansion of the multiple arms of the basket in the infusion catheter causes fissuring of the clot. The net result is that a greater surface area of clot is exposed to both endogenous and exogenously administered lytic agents, thereby promoting clot dissolution.

This study will utilize the Bashir™ Endovascular Catheter and the Bashir Endovascular Catheter with a short basket (BASHIR™ S-B endovascular catheter) to administer catheter directed thrombolysis in patients with submassive PE who have consented and meet all eligibility criteria. The Bashir™ and BASHIR™ S-B endovascular catheters represent a new methodology for localized catheter-based delivery of thrombolytics. The thrombolytic to be used in this study is r-tPA (Genentech Corporation, South San Francisco, USA).

The design of the Bashir Endovascular Catheter with the multiple infusion limbs creating a basket-like formation when expanded, provides an immediate channel for blood flow through the thrombus and a greater surface area in the thrombus for the endogenous and exogenous thrombolytics to take effect, as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent;
2. Age 18 to ≤ 75 years of age;
3. PE symptom duration ≤ 14 days.
4. Filling defect in at least one main or lobar pulmonary artery as determined by contrast enhanced chest CT (CTA);
5. RV/LV diameter ratio ≥ 0.9 by CTA as determined by the investigative site;
6. Willing and able to comply with all study procedures and follow-up.

Exclusion Criteria:

1. CVA or TIA within one (1) year;
2. Head trauma, active intracranial, or intraspinal disease ≤ one (1) year prior to inclusion in the study;
3. Active bleeding from a major organ within one (1) month prior to inclusion in the study;
4. Intracranial condition(s) that may increase the risk of bleeding (e.g., neoplasms, arteriovenous malformations, or aneurysms);
5. Patients with bleeding diatheses;
6. Hematocrit < 30%;
7. Platelets < 100,000/μL;
8. INR > 1.5 if currently on warfarin (Coumadin®);
9. aPTT > 50 seconds in the absence of anticoagulants;
10. Major surgery ≤ 14 days prior to inclusion in the study;
11. Serum creatinine > 2.0mg/dL;
12. Clinician deems high-risk for catastrophic bleeding;
13. History of heparin-induced thrombocytopenia (HIT Syndrome);
14. Pregnancy;
15. SBP < 90 mmHg > 15 minutes within two (2) hours prior to BEC procedure and is not resolved with IV fluids;
16. Any vasopressor support;
17. Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR) during this hospitalization at treating institution and/or referring institution;
18. Evidence of irreversible neurological compromise;
19. Life expectancy < one (1) year;
20. Use of thrombolytics or glycoprotein IIb/IIIa inhibitor within 3 days prior to inclusion in the study;
21. Use of non-vitamin K oral anti-coagulants (NOACs), such as rivaroxaban (Xarelto®), apixaban (Eliquis®), dabigatran (Pradaxa®), edoxaban (Savaysa®) within 48 hours prior to inclusion in the study;
22. Profound bradycardia requiring a temporary pacemaker and/or inotropic support;
23. Previous enrollment in this study;
24. Morbidly obese patient who by the judgement of the investigator is high risk for bleeding;
25. BMI > 45kg/m2;
26. Absolute contraindication to anticoagulation;
27. Uncontrolled hypertension defined as SBP > 175mmHg and / or DBP > 110mmHg with pharmacotherapy within two (2) hours prior to inclusion in the study;
28. Currently participating in another study;
29. Any arterial line placement;
30. Current positive COVID diagnosis, or ≤ 8 weeks negative of COVID, or > 8 weeks from positive COVID test and with current symptoms, or current active viral pneumonia on chest CT scan;
31. In the opinion of the investigator, the subject is not a suitable candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Firth, MD, PhD, MBA, FACC, Principal Investigator — Thrombolex, Inc.
Locations (19):
- United States (19):
  - UCLA, Los Angeles, California
  - Miami Cardiac & Vascular Institute, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Emory, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Loyola University Chicago, Maywood, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - Ascension St. John Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Joseph's Hospital, Liverpool, New York
  - NYU Langone, New York, New York
  - NC Heart, Raleigh, North Carolina
  - Mt Carmel, Columbus, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - Tennova Heart - Turkey Creek, Knoxville, Tennessee
  - CAMC, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bashir R, Foster M, Iskander A, Darki A, Jaber W, Rali PM, Lakhter V, Gandhi R, Klein A, Bhatheja R, Ross C, Natarajan K, Nanjundappa A, Angle JF, Ouriel K, Amoroso NE, Firth BG, Comerota AJ, Piazza G, Rosenfield K, Sista AK. Pharmacomechanical Catheter-Directed Thrombolysis With the Bashir Endovascular Catheter for Acute Pulmonary Embolism: The RESCUE Study. JACC Cardiovasc Interv. 2022 Dec 12;15(23):2427-2436. doi: 10.1016/j.jcin.2022.09.011. Epub 2022 Sep 17. PMID 36121244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BEC Treatment
Started | 109
Completed | 103
Not Completed | 6
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Subjects treated with the Bashir™ Endovascular Catheter
Arm/Group | BEC Treatment
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 64
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: RV/LV Ratio Difference
Description: Observe RV/LV diameter ratio difference between baseline and 48 hours after the completion of r-tPA treatment as measured by contrast enhanced chest CT (CTA).
Time Frame: 48 hours after the completion of r-tPA treatment
Population: Subjects treated with the Bashir™ Endovascular Catheter and had analyzable baseline and 48 hour CTAs.
Measure: Mean (95% Confidence Interval); unit: RV/LV Ratio
Arm/Group | BEC Treatment
Number analyzed (Participants) | 107
RV/LV Ratio
  RV/LV Ratio at Baseline (R0) | 1.66 [1.58 to 1.75]
  RV/LV Ratio within 48 hours of completion of treatment (R48) | 1.10 [1.06 to 1.15]
  Difference (R48-R0) | -0.56 [-0.64 to -0.48]

2. Primary Outcome: Safety: Major Bleeding
Description: Major Bleeding as defined by International Society of Thrombosis and Hemostasis (ISTH), within 72 hours of initiation of r-tPA administration. Bleeding criteria are as follows: Major Bleeding in Non-Surgical Patients
  1. Fatal bleeding; and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; and/or
  3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more or leading to transfusion of two or more units of whole blood or red cells.
Time Frame: Within 72 hours of initiation of r-tPA administration
Population: Subjects treated with the Bashir™ Endovascular Catheter
Measure: Count of Participants; unit: Participants
Arm/Group | BEC Treatment
Number analyzed (Participants) | 109
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was captured from time of the procedure through 30-day follow-up
Arm/Group | BEC Treatment
All-Cause Mortality (participants affected / at risk) | 1/109
Serious Adverse Events (participants affected / at risk) | 7/109
Other Adverse Events (participants affected / at risk) | 18/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEC Treatment (N=109)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alcohol withdrawal syndrom (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEC Treatment (N=109)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Device operational issue (Product Issues) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Haematuria (Vascular disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Arrhythmia (Blood and lymphatic system disorders) | 2 (2)
Fasciculation (Nervous system disorders) | 1 (1)
Abscesses of skin (Infections and infestations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Infarct (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04248868/Prot_SAP_000.pdf